CLINICAL TRIAL: NCT01563276
Title: Postural Instability in Progressive Supranuclear Palsy: Why do Patients With PSP Fall?
Brief Title: Postural Instability in Progressive Supranuclear Palsy
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00007924
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Progressive Supranuclear Palsy; Parkinson's Disease
Keywords: Progressive Supranuclear Palsy; PSP; Falls; Gait; Balance; Parkinson's Disease; PD
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Progressive Supranuclear Palsy: Patients with a diagnosis of probable or possible PSP as defined by the National Institute of Neurological Disorders and Stroke and Society for Progressive Supranuclear Palsy (NINDS-SPSP) diagnostic criteria.
- Parkinson's Disease: Idiopathic PD according to the UK Parkinson"s Disease Society Brain Bank Clinical Diagnosis Criteria (UKPDSBBCDC)
- Healthy Control

SUMMARY:
The purpose of this study is to better understand why individuals with Progressive Supranuclear Palsy (PSP) fall. Understanding the mechanism of gait and balance dysfunction in individuals with PSP may provide us with important early diagnostic tools, allowing for earlier identification of mobility problems and to better evaluate medical therapies aimed at improving motor disability.

The investigators will recruit 10 PSP, 10 PD and 10 healthy controls for the study. All subjects will be asked to come to the OHSU clinic at the Center for Health and Healing for an initial screening visit. They will meet with the primary investigator to conduct a brief interview and physical examination. In addition, they will be asked to answer questions regarding current and past medical illness, how often they fall and what kinds of medications they are on.

Subjects who agree to participate will come to the Oregon Clinical and Translational Research Institute (OCTRI) at OHSU for balance testing. Subjects will be asked to stand or sit on a movable platform with eyes open or closed. Prior to standing on the platform, the investigators will place 6 small sensors on body which are held in place by velcro straps (one on each wrist, ankles, chest and lower back). The platform will then be moved (tilt or slide) while subjects try to keep their balance. During all of the balance tests described above, body movements will be recorded from the sensors on the subjects' body. This data is directly recorded by a computer and analyzed to help us gain better understanding of the subjects' posture and their ability to remain up right.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable or possible PSP as defined by the National Institute of Neurological Disorders and Stroke and Society for Progressive Supranuclear Palsy (NINDS-SPSP) diagnostic criteria.
2. Be able to ambulate and stand unassisted for 5 minutes
3. Be able to cooperate with gait and balance testing
4. Be able to give informed consent.

Exclusion Criteria:

1. Cannot exhibit behavior or have dementia that precludes participation in the protocol
2. Cannot have medical or orthopedic illness that, in the investigator's opinion, would impact the patient's postural control or ability to participate in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OHSU Movement Disorders Clinic Volunteers from the community (Portland, Oregon and surrounding areas)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05-10 (Actual); Study Completion 2013-05-10 (Actual)

PRIMARY OUTCOMES:
Relative contributions of vestibular and visual information to postural control in PSP | Single visit. 2 hours.
  To gage the relative contributions of vestibular and visual information to postural control in PSP we will measure body sway using two different tests (LOS and SOT) while a patient stands on a movable force plate within a movable visual surround.

SECONDARY OUTCOMES:
Postural Response Latencies | Single visit. 2 hours.
  Subjects will stand on a movable platform with a movable visual surround. Subjects will be asked to keep their balance while the platform is translated or roated.
Gait patterns and postural transitions | Single visit. 10 minutes.
  Subjects will be asked to rise from a chair, walk and turn. Ambulatory balance will be measured by a time up and go test (TUG). Six accelerometers will be placed on the subject and will measure parameters including arm swing, number of steps and turn duration.
Perception of vertical and horizontal references | Single visit. 2 hours.
  Subjects will perform two different tasks with their eyes closed while standing and sitting on a force plate that is tilting in the antero-posterior direction. They will perform the following two tasks: 1. Hold a rod parallel to the gravitional vertical 2. Hold a rod perpendicular to the tilting surface so it remains 90 degrees to the surface at all times. Six accelerometers will measure lower and upper body tilt.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Schoneberg, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States